CLINICAL TRIAL: NCT03051984
Title: Skeletal Muscle Atrophy and Dysfunction Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael J. Toth, Ph.D., Associate Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: M16-528; R01AG050305 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthristis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NMES (Experimental): Neuromuscular electrical stimulation (NMES) will be administered for 5 weeks post-TKA in the quadriceps of the surgical leg. Treatment will occur 5 days per week, twice daily for 45 minutes on each occasion.
  Interventions: Device: Neuromuscular electrical stimulation
- Control (No Intervention): No intervention will be administered during the 5 weeks post-TKA in the surgical leg.

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — NMES will be conducted on the quadriceps of the operative leg using a portable stimulation device, starting within 48-72 hrs of surgery. The operative leg will be immobilized at a neutral angle (~30º), with electrodes affixed to the anterior surface of the thigh. Symmetrical, biphasic pulses (400 µs duration at 50 Hz) will be used, with a duty cycle of 25% (10 s on, 30 s off), with patient-selected stimulation intensity to cause visible contractions below pain threshold. NMES sessions will occur 5 d/week, twice daily for 45 min (5 min warm-up) for 5 wks.
  Other Names: NMES
  Arms: NMES

SUMMARY:
Total knee replacement, or arthroplasty, is the final clinical intervention available to relieve pain and functional limitations related to advanced stage knee osteoarthritis. Despite its beneficial effects, the early post-surgical period is characterized by the erosion of lower extremity muscle size and strength that cause further disability and slow functional recovery. While the detrimental effects of this period on muscle are widely recognized, the mechanisms underlying these adaptations are poorly understood and there are currently no widely-accepted clinical interventions to counter them

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is currently the most common elective surgery in the US and will increase in frequency nearly five-fold by 2030 to 3.5 million surgeries annually. This surgery is most prevalent among older adults with advanced knee osteoarthritis (OA) and its increase is explained primarily by growth in this population. Although TKA reliably reduces joint pain, it fails to correct objectively-measured functional disability due, in part, to dramatic declines in lower-extremity neuromuscular function during the early, postsurgical period. These deficits are never fully remediated, remaining for years after surgery and contributing to persistent disability. Despite these detrimental effects of TKA, the fundamental skeletal muscle adaptations that occur in the early, post-surgical period are poorly defined and understudied and there is currently no widely-accepted, evidence-based intervention to counter these changes. To address this clinical problem, the investigators goals in this application are to define the skeletal muscle structural and functional adaptations following TKA at the whole body, tissue, cellular, organellar and molecular levels in humans in an effort to identify factors contributing to functional disability and to assess the utility of neuromuscular electrical stimulation (NMES) to counter post-surgical muscle adaptations at these same anatomic levels. We hypothesize that TKA fails to remediate physical disability in patients, in part, because of the profound skeletal muscle myofilament and mitochondrial loss and dysfunction that develops during the early, post-surgical period. Moreover, the investigators posit that NMES will improve functional recovery following TKA by countering these early skeletal muscle adaptations. To test this model, the investigators will evaluate participants with knee OA prior to and following TKA for skeletal muscle structure and function at multiple anatomic levels, with patients randomized to receive NMES or sham control intervention during the first 5 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic, primary knee osteoarthritis (OA)
* being considered for total knee arthroplasty

Exclusion Criteria:

* knee OA secondary to inflammatory/autoimmune disease
* untreated/uncontrolled hypertension, diabetes or thyroid disease
* chronic heart failure, actively-treated malignancy, exercise-limiting peripheral vascular disease, stroke or neuromuscular disease
* body mass index >38 kg/m2
* lower extremity blood clot or known coagulopathies
* implanted pacemaker/ICD

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on January 1, 2017, and ended on January 13, 2022. Volunteers undergoing assessment for TKA were screened from the Adult Reconstruction Service of our Department of Orthopedics and Rehabilitation and local private practices.
Groups:
- Experimental: NMES: Volunteers randomized to this arm/group will receive neuromuscular electrical stimulation (NMES) for 5 weeks after total knee arthroplasty (TKA)
- Experimental: Control: Patients randomized to this arm/group will not receive any experimental intervention, but will receive standard of care.
Period: Overall Study
Arm/Group | Experimental: NMES | Experimental: Control
Started | 11 | 12
Completed | 10 | 11
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: NMES | Experimental: Control | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (7.1) | 64.8 (6.5) | 64.0 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cross-sectional Area (CSA) of Muscle Fibers
Description: CSA of skeletal muscle fibers via myosin heavy chain (MHC) immunohistochemistry
Time Frame: Baseline and 5-weeks post-TKA surgery
Population: Mixed model analysis statistically adjusted for baseline value and sex
Measure: Least Squares Mean (Standard Error); unit: micron squared
Arm/Group | Experimental: NMES | Experimental: Control
Number analyzed (Participants) | 10 | 10
micron squared
  MHC I fiber cross-sectional area - Baseline | 2680 (113) | 2377 (86)
  MHC I fiber cross sectional area - 5-week post-surgery | 2028 (83) | 1882 (68)
  MHC IIA fiber cross sectional area - Baseline | 2039 (183) | 1971 (155)
  MHC IIA fiber cross sectional area - 5-week post-surgery | 1623 (145) | 1389 (109)

2. Primary Outcome: Intermyofibrillar Mitochondrial Content
Description: Fractional area of intermyofibrillar (IMF) mitochondria via electron microscopy
Time Frame: Baseline and 5-weeks post-TKA surgery
Population: Mixed model analysis adjusting for baseline value and sex
Measure: Least Squares Mean (Standard Error); unit: percent area
Arm/Group | NMES | Control
Number analyzed (Participants) | 10 | 10
percent area
  IMF mitochondria fractional area - Baseline | 2.36 (0.20) | 2.34 (0.20)
  IMF mitochondria fractional area - 5-week post-surgery | 2.1 (0.20) | 1.7 (0.20)

3. Primary Outcome: Maximal Calcium-activated Tension Single Muscle Fiber Tension
Description: Tension (force per unit muscle fiber cross-sectional area) from segments of chemically-skinned single human muscle fibers assessed under maximal calcium-activated condition, with muscle fiber type determined post-measurement by gel electrophoresis
Time Frame: Baseline and 5-weeks post-TKA surgery
Population: Mixed model analysis adjusting for baseline value and sex.
Measure: Least Squares Mean (Standard Error); unit: milliNewtons per millimiter squared
Arm/Group | Experimental: NMES | Experimental: Control
Number analyzed (Participants) | 8 | 8
milliNewtons per millimiter squared
  MHC I tension - Baseline | 114 (5) | 111 (5)
  MHC I tension - 5-week post-surgery | 112 (5) | 103 (5)
  MHC IIA tension - Baseline | 173 (5) | 175 (6)
  MHC IIA tension - 5-week post-surgery | 132 (6) | 107 (8)

4. Secondary Outcome: Physical Activity Level
Description: Physical activity will be assessed by accelerometry.
Time Frame: Baseline and 5-weeks post-TKA surgery
Population: Analysis of variance. Note that one patient in the control group did not complete accelerometry assessments.
Measure: Mean (Standard Error); unit: steps per day
Arm/Group | Experimental: NMES | Experimental: Control
Number analyzed (Participants) | 10 | 10
steps per day
  Step counts - Baseline | 4167 (688) | 4767 (691)
  Step counts - 5-week post-surgery | 2088 (588) | 2500 (587)

5. Secondary Outcome: Quadriceps Muscle Cross-sectional Area
Description: Quadriceps muscle cross-sectional area will be assessed by computed tomography at the mid-thigh on both surgical and non-surgical non-surgical legs.
Time Frame: Baseline and 5-weeks post-TKA surgery
Population: Mixed model analysis with control for baseline value and sex
Measure: Mean (Standard Error); unit: centimeters squared
Arm/Group | Experimental: NMES | Experimental: Control
Number analyzed (Participants) | 10 | 11
centimeters squared
  Surgical Quadriceps cross-sectional area - Baseline | 45.5 (3.0) | 38.8 (3.1)
  Surgical Quadriceps cross-sectional area - 5-week post-surgery | 38.3 (3.3) | 33.8 (2.7)
  Non-surgical Quadriceps cross-sectional area - Baseline | 52.0 (3.3) | 46.0 (4.5)
  Non-surgical Quadriceps cross-sectional area - 5-week post-surgery | 48.7 (3.6) | 44.9 (3.9)

6. Secondary Outcome: Short Physical Performance Battery
Description: Physical functional assessment based on 2 lower extremity activities (5-time sit-to-stand, 4-m gait speed) and standing balance (side-side, tandem, semi-tandem) based on time or repetitions (0-4 score) with a minimum score of 0 and a maximal score of 12. Each activity is scored from 0 to 4 based on the level of performance (with higher values indicating better physical function and lower values indicating increasing levels of disability). The scores from the 3 activities are summed to give the total score, which is what is reported. Higher total score values indicate higher levels of physical function (more healthy), whereas lower values indicate increasing levels of physical disability/frailty.
Time Frame: Baseline and 5-weeks post-TKA surgery
Population: Analysis of variance.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Experimental: NMES | Experimental: Control
Number analyzed (Participants) | 10 | 11
Scores on a scale
  Short Physical Performance - Baseline | 9.36 (0.56) | 9.80 (0.61)
  Short Physical Performance Battery - 5-week post-surgery | 10.45 (0.53) | 10.10 (0.55)

7. Secondary Outcome: Knee Extensor Muscle Strength
Description: Knee extensor isometric peak torque assessed by dynamometry on the surgical leg.
Time Frame: Baseline and 5-weeks post-TKA surgery
Population: Analysis of variance model. Note that n=9 for surgical leg isokinetic peak torque in one NMES volunteer because knee pain prevented completing of strength testing protocol.
Measure: Mean (Standard Error); unit: Newton meter
Arm/Group | Experimental: NMES | Experimental: Control
Number analyzed (Participants) | 9 | 11
Newton meter
  Surgical Isometric peak torque - Baseline | 113.0 (14.5) | 94.7 (9.8)
  Surgical Isometric peak torque - 5-week post-surgery | 65.8 (6.9) | 65.7 (6.9)
  Surgical Isokinetic peak torque - Baseline | 89.9 (9.6) | 58.9 (9.6)
  Surgical Isokinetic peak torque - 5-week post-surgery | 53.3 (4.2) | 42.5 (3.9)

8. Secondary Outcome: 30-second Sit-to-stand Test
Description: Number of repetitions that an individual can complete the sit-to-stand transition in 30 seconds
Time Frame: Assessed at baseline and 5 weeks post-surgery
Population: Analysis of variance model.
Measure: Mean (Standard Error); unit: repetitions
Arm/Group | Experimental: NMES | Experimental: Control
Number analyzed (Participants) | 10 | 11
repetitions
  30-s sit-to-stand - Baseline | 10.45 (0.97) | 11.78 (1.39)
  30-s sit-to-stand - Post-surgery | 10.55 (0.59) | 12.56 (1.22)

ADVERSE EVENTS:
Time Frame: Enrollment to end of follow-up, an average of 5 weeks
Arm/Group | Experimental: NMES | Experimental: Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: NMES (N=10) | Experimental: Control (N=11)
Low-dose x-ray exposure outside of protocol specified exposure. (General disorders) | 1 | 0 — Patient exposed to additional low-dose x-ray during dual energy x-ray absorptiometry (DEXA) scan due to error in DEXA scanner software. Mild, unrelated to intervention.
Excessive bleeding during muscle biopsy procedure. (Musculoskeletal and connective tissue disorders) | 0 | 1 — Excessive bleeding after completion of skeletal muscle biopsy. Mild, unrelated to intervention.
Tinea pedis (Skin and subcutaneous tissue disorders) | 0 | 1 — Tinea pedis. Mild, unrelated to intervention or participation in study.

LIMITATIONS AND CAVEATS:
Recruitment for the study was curtailed by the COVID-19 pandemic and its associated research closures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03051984/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03051984/SAP_001.pdf